CLINICAL TRIAL: NCT04508972
Title: Voice-based Identification of Clinical Features Requiring Emergent Action in Patients With Suspected COVID-19 Infection (VOICE-COVID) I and II Study
Brief Title: The VOICE-COVID-19
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Amazon Web Services (AWS) Canada (Unknown)
Responsible Party: Principal Investigator, Abhinav Sharma, Cardiologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2020-6583
Record Dates: First submitted 2020-08-10; First posted 2020-08-11 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Covid19
Keywords: COVID-19; Alexa Device; Voice-based technologies; Screening; Safety
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Alexa Amazon — To test the use of the Amazon Alexa device as a tool to conduct screening of employees and patients at the point of entry into the Heart Failure (HF) Clinic of the McGill University Health Center.

SUMMARY:
The VOICE-COVID study will evaluate the concordance of screening for symptoms of COVID-19 using a voice based device (Amazon Alexa) compared to manual screening by a study coordinator for individuals entering the Cardiology/Heart Failure clinic at the McGill University Health Centre.

DETAILED DESCRIPTION:
This study is an open-label, prospective, cross-over randomized study.

VOICE-COVID I: All individuals entering the Heart Failure (HF) Clinic of the McGill University Health Center will be asked to participate. A poster with instructions to ask the participants (employees or patients) to speak with the Amazon Alexa device. The participant will remain 6 feet away from the device. The Amazon Alexa will ask the survey questions. A study coordinator will then ask the same questions along with some additional questions about Amazon Alexa usability. VOICE-COVID II: A second cohort of 52 people will be then randomized to be screened for symptoms of COVID-19 with an Amazon Alexa or a coordinator. We will study the correlation between the Alexa response and the response to the study coordinator using K-squared statistic tests and screening question concordance.

ELIGIBILITY:
Inclusion Criteria:

* Adults >=18 yrs who is entering the HF clinic
* Speaks either English or French

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any employees or patients entering the Heart Failure clinic at the McGill University Health Center
Sampling Method: Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Correlation between data captured using Amazon Alexa compared to manual (human) collected data. | Day 1
  Determine the ability of the Amazon Alexa device to properly capture answers from participants and correlate with the answers retrieved by the study coordinator.

OTHER OUTCOMES:
Self reported Likert scale on comfort in using the Amazon Alexa device | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Abhinav Sharma, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Muhc-Rimuhc, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We aim to disseminate these results through publications in peer review journals and submission to conferences. Currently, many conferences are converting into a virtual format which would enable our results to be disseminated over a wide audience.

REFERENCES:
- [Derived] Marques P, Emami A, Zhang G, Lopes RD, Razaghizad A, Avram R, Sharma A. Impact of age and comorbid heart failure on the utility of smart voice-assistant devices. Eur Heart J Digit Health. 2024 Feb 16;5(3):389-393. doi: 10.1093/ehjdh/ztae012. eCollection 2024 May. PMID 38774370
- [Derived] Sharma A, Marques P, Zhang G, Oulousian E, Chung SH, Ganni E, Lopes RD, Razaghizad A, Avram R. Voice-assisted Artificial Intelligence-enabled Screening for Severe Acute Respiratory Syndrome Coronavirus 2 Exposure in Cardiovascular Clinics: Primary Results of the VOICE-COVID-19-II Randomized Trial. J Card Fail. 2023 Oct;29(10):1456-1460. doi: 10.1016/j.cardfail.2023.05.004. Epub 2023 May 22. PMID 37224994
- [Derived] Oulousian E, Chung SH, Ganni E, Razaghizad A, Zhang G, Avram R, Sharma A. Voice-Based Screening for SARS-CoV-2 Exposure in Cardiovascular Clinics (VOICE-COVID-19-II): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Jan 31;12:e41209. doi: 10.2196/41209. PMID 36719720
- [Derived] Sharma A, Oulousian E, Ni J, Lopes R, Cheng MP, Label J, Henriques F, Lighter C, Giannetti N, Avram R. Voice-based screening for SARS-CoV-2 exposure in cardiovascular clinics. Eur Heart J Digit Health. 2021 Jun 16;2(3):521-527. doi: 10.1093/ehjdh/ztab055. eCollection 2021 Sep. PMID 36713601